CLINICAL TRIAL: NCT03643549
Title: Bortezomib Sensitization of Recurrent Grade-4 Glioma With Unmethylated MGMT Promoter to Temozolomide Phase 1B/II Study
Brief Title: Bortezomib and Temozolomide in Recurrent Grade-4 Glioma Unmethylated MGMT Promoter (BORTEM-17)
Acronym: BORTEM-17
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Oslo University Hospital (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other); University of Bergen (Other); University of Bonn (Other); University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017/2084
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Glioblastoma
Keywords: Temozolomide; Bortezomib; Recurrent disease
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Bortezomib

STUDY DESIGN:
Intervention Model Description: Botezomib 1.3mg/m2 administered IV on days 1, 4, 7, during each 4-week chemotherapy cycle with per oral Temozolomide at three dose levels: 150 mg/m2, 175 mg/m2 and 200mg/m2 5 days/week every 4 weeks starting on day 3 until disease progression and/or unacceptable toxicity. Study group will be compared to historical controls on conventional management
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bortezomib and Temozolomide (Experimental): Botezomib 1.3 mg/m2 administered IV on days 1, 4, 7, during each 4-week chemotherapy cycle with per oral Temozolomide at three dose levels: 150 mg/m2, 175 mg/m2 and 200mg/m2 5 days/week every 4 weeks starting on day 3.
  Interventions: Drug: Bortezomib and Temozolomide Phase IB; Drug: Bortezomib and Temozolomide Phase II

INTERVENTIONS:
Drug: Bortezomib and Temozolomide Phase IB — In the Phase IB of the study the following dose escalation of TMZ will be performed: The first cohort of 3 patients will receive 150 mg/m2 of IMP (TMZ) for 5 days q4w. If one patient in this cohort develops a dose limiting toxicity, another cohort of 3 patients will be treated at the same dose level until 2 or more patients in the group of 3-6 develop DLT.
Drug: Bortezomib and Temozolomide Phase II — The patientes will be treated with the maximum recommended starting dose of Temozolomide and Bortezomib established in the IB phase of the study

SUMMARY:
This phase IB/II trial is designed to investigate the safety and survival benefits for patients with recurrent grade-4 with unmethylated MGMT promoter treated with Bortezomib and Temozolomide in a specific schedule.

DETAILED DESCRIPTION:
Patients harbouring tumours with functional O6 methylguanine DNA methyltransferase (MGMT) DNA repair enzyme efficiently repair the DNA damage inflicted by Temozolomide and gain limited benefit from this chemotherapy. Bortezomib depletes the MGMT enzyme, restoring the tumour´s susceptibility to Temozolomide, if the chemotherapy is administered in the precise schedule when the MGMT enzyme is depleted. Additionally, Bortezomib inhibits the growth of tumour cells by blocking autophagy flux. Temozolomide causes genotoxic stress in cancer cells that in turn respond by inducing protective processes such as autophagy. If both autophagy and MGMT DNA repair enzyme are blocked a priori, the efficacy of Temozolomide will be enhanced. Thus, pre-treating the tumour with Bortezomib prior to administration of Temozolomide leads to DNA repair enzyme depletion and blockade of autophagy-induced survival signals. The combined effect will sensitize the tumour to therapy, improve chemotherapy efficacy and prolong patient survival outcomes.

Hypothesis: Pretreatment with Bortezomib administered prior to Temozolomide will sensitize recurrent GBM with unmethylated MGMT promoter to standard TMZ in palliative setting.

Objective:

* Assessment of safety and tolerability of Bortezomib administered with Temozolomide.
* Determining the optimal dose of TMZ, when administered as combination therapy
* Estimate the progression free survival (PFS) and overall survival (OS) of patients with recurrent or progressed glioblastoma after pre-treatment with Bortezomib prior to combination with Temozolomide.

Key secondary objectives

* Tumour response to the therapy assessed by RANO and NANO criteria
* Determine physiological, molecular and biochemical changes in blood and tumour tissue that correlate with treatment responses.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy > 8 weeks
* Histologically confirmed intracranial glioblastoma (GBM), with MGMT unmethylated promoter
* Must submit an unstained paraffin block and/ or cryopreserved tumour tissue from surgical procedure
* Radiologically (MRI) confirmed tumour relapse/progression ≥ 12 weeks since completed radiotherapy
* Measurable recurrent tumor
* Tumor not available for radio-surgery
* If previously treated with gammaknife, at least one evaluable lesion outside the irradiated area is required, unless the time after the radiosurgery is 12 weeks or more
* Written informed consent for study participation and tumour, blood sample collection obtained before performance of any study related procedure.
* Karnofsky performance status ≥ 70
* WBC ≥ 3,000/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* Bilirubin < 2.5 times upper limit of normal (ULN)
* serum aspartate aminotransferase (AST) < 2.5 times ULN
* Estimated GFR ≥ 60 mL/minute
* Serum sodium > 130 mmol/L
* Serum potassium level within normal limit
* Stable or reduced doses of corticosteroids for at least 1 week prior to enrolment
* Negative pregnancy test no longer than 14 days prior to enrollment
* Fertile patients and female partners with child bearing potential of male patients must use adequate contraception
* Patients on EIAED must be transitioned to non-EAIED for ≥ 2 weeks
* Unfractionated and/or low molecular weight heparin allowed
* Patients previously treated with neurosurgery er eligible for the study

Exclusion Criteria:

* Hypersensitivity to Bortezomib, boron, or mannitol
* Any contraindications for use of temozolomide
* Peripheral neuropathy ≥ grade 2
* Previous treatment with bevacizumab or lomustine alone or as a combination therapy for ralapsed glioblastoma (PCV as primary treatment of low grade glioma, before development of glioblastoma, is allowed)
* Myocardial infarction within the past 6 months
* NYHA class III or IV heart failure
* Uncontrolled angina
* Severe uncontrolled ventricular arrhythmias
* Electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Known heart failure
* Serious medical or psychiatric illness that would interfere with the study participation including, but not limited to, any of the following:
* Ongoing or active infection requiring IV antibiotics
* Psychiatric illness and/or social situations that would limit compliance with study requirements
* Disorders associated with a significant immunocompromised state (e.g., HIV, systemic lupus erythematosus)
* History of stroke within the past 6 months
* Other malignancy within the past 3 years except completely resected basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy (i.e., cervical cancer), or low-risk prostate cancer after curative therapy
* Significant medical illness that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* Disease that will obscure toxicity or dangerously alter the drug metabolism
* Viral hepatitis (HBV surface antigen positive) or active hepatitis C infection
* Other investigational drugs must be stopped at least 12 weeks prior to therapy or treatment failure under other experimental therapy must be confirmed before study entry. If progression during other experimental therapy is confirmed, the time interval between previous treatment and BORTEM-17 may be reduced to 4 weeks
* Concurrent inducers of CYP450 3A4 (e.g., enzyme-inducing anti-epileptic drugs [EIAED])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bortezomib-Temozolomide Maximum tolerated dose | 6 months
  En intra- and inter-patient dose escalation period of TMZ administered after Bortezomib
Overall survival | 1 year
  Overall survival at 1 year
Progression free survival | 6 months
  Progression free survival at 6 months
Time to progression | 4 years
  Median time

SECONDARY OUTCOMES:
Biomarkers of treatment response | 4 years
  Identification of novel tumor biomarkers by determining physiological, molecular and biochemical changes in blood and tumor tissue that correlate with treatment responses
Tumour responses | 4 years
  Assessed by contrast enhanced MRI according to RANO criteria
Clinical response | 4 years
  Assessment of the neurologic status according to NANO criteria
Toxicity assessment | 4 years
  SAE, all grades hematologic and non hematologic toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Goplen, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo

REFERENCES:
- [Derived] Rahman MA, Brekke J, Arnesen V, Hannisdal MH, Navarro AG, Waha A, Herfindal L, Rygh CB, Bratland E, Brandal P, Haasz J, Oltedal L, Miletic H, Lundervold A, Lie SA, Goplen D, Chekenya M. Sequential bortezomib and temozolomide treatment promotes immunological responses in glioblastoma patients with positive clinical outcomes: A phase 1B study. Immun Inflamm Dis. 2020 Sep;8(3):342-359. doi: 10.1002/iid3.315. Epub 2020 Jun 24. PMID 32578964